CLINICAL TRIAL: NCT03061019
Title: Comparison of Two Oral Myofunctional Reeducation Methods for Children With Obstructive Sleep Apnea Before Adenotonsillectomy : a Randomized Controlled Trial.
Brief Title: Comparison of Two Oral Myofunctional Reeducation Methods for Children With Obstructive Sleep Apnea
Acronym: PERSIST-B
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: a RCT was started
Sponsor: Université de Montréal (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Nelly Huynh, Professor, PhD, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1297
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: child; myofunctional therapy; adenotonsillectomy; randomized controlled trial
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Myofunctional Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofunctional Oral Exercices (Active Comparator): Parents and participants of this group will receive instructions for nasal and oral myo-functional exercises, to perform at home each day, for 5 to 10 minutes. A booklet (measure of adherence) and an Phone application for Android/Apple with descriptions/videos of those exercices will be given to them. These exercises will include nasal hygiene procedures, nasal cartilage exercices, lingual posture rehabilitation exercises, lip tone enhancement exercises, and swallowing rehabilitation exercises.
  Interventions: Procedure: Oral Myofunctional Therapy with exercices
- Soft Oral Appliance (Experimental): Parents and participants will be instructed in wearing the soft/flexible oral appliance and how to perform nasal hygiene in order to better tolerate the device. The oral appliance comes in several sizes, adapted to the age of the child; it is constructed in a soft elastomer material, in a position of slight propulsion and opening of the mandible to help clear the pharynx. It has a ramp to guide the tongue in a good position, a labial screen to stretch the labial strap and prevent the tongue from protruding between front teeth.
  Interventions: Procedure: Oral Myofunctional Therapy with soft oral appliance
- Control Group (No Intervention): Parents and Participants of this group will be reminded the nasal hygiene procedures (application of saline in each nostril three times a day), and given a diary to report daily use.

INTERVENTIONS:
Procedure: Oral Myofunctional Therapy with exercices — Oral-Motor training of oral muscles (tongue, lips) associated with nasal hygiene with daily repetition of exercices and parental support.
  Other Names: Oral reeducation
  Arms: Myofunctional Oral Exercices
Procedure: Oral Myofunctional Therapy with soft oral appliance — Ora-Motor training of oral muscles (tongue, lips) associated with nasal hygiene, with reduced parental support.
  Other Names: Oral Trainer
  Arms: Soft Oral Appliance

SUMMARY:
Myofunctional therapy has been shown to be effectively reduce symptoms of paediatric sleep apnea. As the effectiveness of reeducation relies on parental involvement and child's compliance, the investigator's research question was to evaluate two methods of myofunctional therapy (daily oral exercices versus a flexible oral appliance, both in combination with nasal hygiene), compared to nasal hygiene alone (control group).

DETAILED DESCRIPTION:
Introduction: Paediatric Obstructive Sleep Apnea (OSA) is a multifactorial condition, associated with significant comorbidities, affecting cardiovascular health, cognitive development and quality of life. Its main cause is adenotonsillar hypertrophy, but some co-factors such as obesity, orofacial dysfunctions and craniofacial abnormalities contribute to the severity of symptoms or their persistance after adeno-tonsillectomy.

Aim : Myofunctional therapy has been shown to reduce Apnea-Hyponea indexes (AHI) of children, and can serve as an adjunct to other therapies, but the level of compliance is a limiting factor. The investigator's aim is to evaluate two methods of oral reeducation in a group a children scheduled for adeno-tonsillectomy (in association with nasal hygiene) and to compare them with nasal hygiene alone (control group).

Methods : The design of the study is a randomized Controlled Trial, enrolling 60 children with significant obstructive sleep apnea and divided into 3 groups : Group 1 following daily oral exercises (+nasal hygiene), Group 2 using of a flexible oral appliance during quiet activities and sleep (+nasal hygiene), and Group 3 using nasal hygiene alone (control group). The objective assessment of sleep parameters is performed at home using an ambulatory device (AHI, desaturation index, minimal oxygen saturation, flow limitation, snoring), before and after therapy, in a 3 months interval. An orthodontic and craniofacial assessment, the examination of orofacial functions and tongue/lip strength measurements (IOPI system), as well as quality of life questionnaires (OSA-18) are also performed on participants, before and after therapy.

ELIGIBILITY:
Inclusion Criteria: participants must:

* present signs of obstructive sleep apnea: snoring, apnea / respiratory pauses audible by the entourage (objectivized by a score, to the hierarchical questionnaire of severity of Spruyt and Gozal, greater than or equal to 2,72- This questionnaire comprises six Questions and has a good sensitivity (60%) and specificity (82%) in screening for pediatric sleep apnea.
* be programmed for adenoidectomy, tonsillectomy or adeno-tonsillectomy within 3 months (or more).

Exclusion Criteria: participants should not:

* present with a craniofacial syndrome nor a severe medical condition with complex medical management,
* present with an abnormality of the neuromuscular tone (such as Duchenne myopathy or cerebral palsy)
* receive orthodontic therapy during the study
* have a class III malocclusion (mandibular prognathy type), for which a propulsion oral appliance is contraindicated because it may aggravate mandibular prominence. Maxillary deficiency is not a exclusion criterion.
* A non-nutritive oral habit such as digital sucking (or pacifier) that persists because it interferes with oral reeducation, and is a contraindication to orthodontic treatments. Children who have recently stopped such a habit may be included in the study.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Sleep Parameters Changes : Apnea Hypopnea Index (AHI) | Baseline and 3 months
  Full Night Polygraph using an ambulatory device Type III (cardio-respiratory); measurement of the index of apnea and hypopnea/ in relation to total sleep time, according the American Association of Sleep Medicine (AASM) recommandations for children.
Sleep Parameters Changes : Oxygen desaturation index (ODI) | Baseline and 3 months
  Full Night Polygraph using an ambulatory device Type III (cardio-respiratory); measurement of the index of oxygen desaturation per hour/ in relation to total sleep time, according the American Association of Sleep Medicine (AASM) recommandations for children (oximetry).
Sleep Parameters Changes : Flow Limitation index | Baseline and 3 months
  Full Night Polygraph using an ambulatory device Type III (cardio-respiratory); measurement of flow limitations per hour , in relation to total sleep time, according the American Association of Sleep Medicine (AASM) recommandations for children (nasal canula or thermistance).

SECONDARY OUTCOMES:
Oral muscles strength | Baseline and 3 months
  Lip and Tongue strength and endurance measurement with the IOPI measurement system: Measurement of Anterior and Posterior tongue elevation strength (kPa), Lip Seal strength (kPa)
Nasal Resistance | Baseline and 3 months
  Nasal resistance measurements with a anterior rhino-manometry : effective resistance left nostril (expiration, inspiration), effective resistance right nostril Pa/cm3/s during expiration, inspiration) ,total breath resistance (Pa/cm3/s during expiration, inspiration), vertex resistance right, vertex resistance left (Pa/cm3/s during inspiration, expiration).
Quality of Life | Baseline and 3 months
  OSA 18 Questionnaire, consisting of a 18-items score and Visual Analog scale (from 0 to 10), filled by parents.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Huynh, PhD, Principal Investigator — Université de Montréal, Montréal, Québec, Canada; Marie-Claude Quintal, MD, Principal Investigator — Hôpital Sainte-Justine, Montréal, QC, Canada
Locations (1):
- CHU Sainte Justine, Université de Montréal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Undecided